CLINICAL TRIAL: NCT06596759
Title: Diaphragmatic Breathing for the Treatment of Bloating and Distension: a Prospective Pilot Study
Brief Title: Diaphragmatic Breathing for the Treatment of Bloating and Distension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brian Lacy, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-002905
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Bloating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diaphragmatic Breathing (Experimental): Patients will complete the Mayo Bloating Questionnaire (MBQ) before referral to a physical therapist for in diaphragmatic breathing (DB) techniques over a 30-minute session. The patient will be instructed to complete 5-10 minutes of diaphragmatic breathing twice a day for a period of 4 weeks. At the end of the 4-week follow up period, patients will repeat the MBQ and self-report their adherence to daily diaphragmatic breathing.
  Interventions: Behavioral: Diaphragmatic Breathing

INTERVENTIONS:
Behavioral: Diaphragmatic Breathing — REDCap will be used to administer the Mayo Bloating Questionnaire (MBQ) and collect self-reported compliance to diaphragmatic breathing (DB) exercises over a 4 week follow up period. After completion of the MBQ, the patient will be taught DB techniques by an individual physical therapist face to face over a 30-minute session. The patient will be instructed to complete 5-10 minutes of diaphragmatic breathing twice a day for a period of 4 weeks. Patients will receive a telephone call and electronic health record portal message to check progress and answer any questions. At the end of the 4-week follow up period, patients will repeat the MBQ and self-report their adherence to daily diaphragmatic breathing. The questionnaire will include prompts investigating perceived side effects and attitudes towards therapy, willingness to perform DB therapy, likelihood to attempt self-guided DB in the future, and if the participant would recommend the therapy to a friend.

SUMMARY:
The purpose of this study is to evaluate the efficacy of diaphragmatic breathing using the validated Mayo Bloating Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Referred for breath testing for the indication of bloating.

Exclusion Criteria:

* Not referred for breath testing for the indication of bloating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Mayo Bloating Questionnaire (MBQ) score | Baseline, 4 weeks
  The Mayo Bloating Questionnaire is a 45-item questionnaire developed to measure the multiple symptom components of bloating and distension.

CONTACTS AND LOCATIONS:
Overall Officials: Brian E Lacy, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No